CLINICAL TRIAL: NCT02201940
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Sofosbuvir/GS-5816 Fixed Dose Combination for 12 Weeks in Subjects With Chronic HCV
Brief Title: Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks in Adults With Chronic HCV Infection
Acronym: ASTRAL-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-342-1138; 2014-001683-35 (EudraCT Number)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2016-07

CONDITIONS: Hepatitis C Virus Infection
Keywords: Sofosbuvir; SOF/VEL; Velpatasvir; Hepatitis C; HCV; cirrhosis
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOF/VEL (Experimental): SOF/VEL for 12 weeks
  Interventions: Drug: SOF/VEL
- Placebo (Placebo Comparator): SOF/VEL placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily
  Other Names: Epclusa®; GS-7977/GS-5816
  Arms: SOF/VEL
Drug: Placebo — Tablet administered orally once daily
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of sofosbuvir/velpatasvir (SOF/VEL) fixed dose combination (FDC) for 12 weeks in adults with chronic genotype 1, 2, 4, 5, or 6 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA ≥ 10^4 IU/mL at screening
* HCV genotype 1, 2, 4, 5, 6, or indeterminate assessed at screening by the central laboratory
* Chronic HCV infection (≥ 6 months) documented by prior medical history or liver biopsy
* Classification as treatment naive or treatment experienced
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception

Exclusion Criteria:

* Current or prior history of clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with treatment, assessment, or compliance with the protocol; individuals currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
* Screening ECG with clinically significant abnormalities
* Laboratory results outside of acceptable ranges at Screening
* Prior exposure to SOF or other nucleotide analogue HCV NS5B inhibitor or any HCV NS5A inhibitor
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McNally, PhD, Study Director — Gilead Sciences
Locations (69):
- United States (30):
  - Little Rock, Arkansas
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - New York, New York
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Nashville, Tennessee
  - San Antonio, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
- Belgium (3):
  - Antwerp
  - Brussels
  - Kortrijk
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Montreal, Quebec
  - Toronto
- Hong Kong, China
- France (11):
  - Clermont-Ferrand
  - Clichy
  - Créteil
  - Lille
  - Limoges
  - Lyon
  - Marseille
  - Paris
  - Pessac
  - Toulouse
  - Villejuif
- Germany (8):
  - Frankfurt am Main, Hessin
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Hufelandstr, North Rhine-Westphalia
  - Berlin
  - Hamburg
  - Hanover
  - München
- Italy (2):
  - San Giovanni Rotondo, Foggia
  - Florence
- San Juan, Puerto Rico
- United Kingdom (7):
  - Plymouth, Devon
  - Portsmouth, Hampshire
  - Glasgow
  - London
  - Manchester
  - Nottingham
  - Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Asselah T, Charlton M, Feld J, Foster GR, Mcnally J, Brainard DM, et al. The ASTRAL Studies: Evaluation of SOF/GS-5816 Single Tablet Regimen for the Treatment of Genotype 1-6 HCV Infection [Poster P1332]. J Hepatol 2015;62:S855-S6.
- [Result] Feld JJ, Jacobson IM, Hezode C, Asselah T, Ruane PJ, Gruener N, Abergel A, Mangia A, Lai CL, Chan HL, Mazzotta F, Moreno C, Yoshida E, Shafran SD, Towner WJ, Tran TT, McNally J, Osinusi A, Svarovskaia E, Zhu Y, Brainard DM, McHutchison JG, Agarwal K, Zeuzem S; ASTRAL-1 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 1, 2, 4, 5, and 6 Infection. N Engl J Med. 2015 Dec 31;373(27):2599-607. doi: 10.1056/NEJMoa1512610. Epub 2015 Nov 16. PMID 26571066
- [Result] Feld JJ, Agarwal K, Hezode C, Asselah T, Ruane PJ, Gruener N, et al. A Phase 3 Double-Blind Placebo-Controlled Evaluation of Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks in Naive and Experienced Genotype 1, 2, 4, 5, 6 HCV Infected Patients with and without Cirrhosis: Results of the ASTRAL-1 Study. J Hepatol 2015;62(6) Suppl:1379A-1380A.
- [Derived] Jacobson IM, Bourgeois S, Mathurin P, Thuluvath P, Ryder SD, Gerken G, Hernandez C, Vanstraelen K, Scherbakovsky S, Osinusi A, Tedesco D, Foster GR. The tolerability of sofosbuvir/velpatasvir for 12 weeks in patients treated in the ASTRAL 1, 2 and 3 studies: A pooled safety analysis. J Viral Hepat. 2023 May;30(5):448-454. doi: 10.1111/jvh.13814. Epub 2023 Mar 2. PMID 36740893
- [Derived] Younossi ZM, Stepanova M, Feld J, Zeuzem S, Sulkowski M, Foster GR, Mangia A, Charlton M, O'Leary JG, Curry MP, Nader F, Henry L, Hunt S. Sofosbuvir and Velpatasvir Combination Improves Patient-reported Outcomes for Patients With HCV Infection, Without or With Compensated or Decompensated Cirrhosis. Clin Gastroenterol Hepatol. 2017 Mar;15(3):421-430.e6. doi: 10.1016/j.cgh.2016.10.037. Epub 2016 Nov 12. PMID 27847279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Canada, Europe, and Asia. The first participant was screened on 18 July 2014. The last study visit occurred on 23 September 2015.
Pre-assignment Details: 847 participants were screened.
Groups:
- SOF/VEL: Sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet administered orally once daily for 12 weeks
- Placebo: SOF/VEL placebo tablet administered orally once daily for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL | Placebo
Started | 625 | 116
Completed | 613 | 0
Not Completed | 12 | 116
Not completed — Randomized/Enrolled but Never Treated | 1 | 0
Not completed — Lack of Efficacy | 2 | 113
Not completed — Lost to Follow-up | 5 | 0
Not completed — Withdrew Consent | 2 | 1
Not completed — Investigator's Discretion | 1 | 1
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug.
Groups:
- SOF/VEL: SOF/VEL (400/100 mg) FDC tablet administered orally once daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL | Placebo | Total
Number analyzed (Participants) | 624 | 116 | 740
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10.9) | 53 (10.4) | 54 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 48 | 298
  Male | 374 | 68 | 442
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 5 | 36
  Not Hispanic or Latino | 589 | 111 | 700
  Unknown or Not Reported | 4 | 0 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 52 | 12 | 64
  White | 493 | 89 | 582
  Asian | 62 | 11 | 73
  American Indian/ Alaska Native | 7 | 0 | 7
  Hawaiian or Pacific Islander | 1 | 1 | 2
  Other | 6 | 3 | 9
  Not Disclosed | 3 | 0 | 3
Region of Enrollment [Number; unit: participants] — All randomized participants were analyzed for Region of Enrollment (N = 741).
  participants
    Canada | 55 | 7 | 62
    Belgium | 40 | 5 | 45
    United States | 234 | 45 | 279
    China | 19 | 4 | 23
    Italy | 16 | 2 | 18
    United Kingdom | 91 | 13 | 104
    France | 126 | 32 | 158
    Germany | 44 | 8 | 52
Cirrhosis Status [Number; unit: participants]
  Present | 121 | 21 | 142
  Absent | 501 | 95 | 596
  Missing | 2 | 0 | 2
HCV Genotype [Number; unit: participants]
  Genotype 1 | 328 | 65 | 393
  Genotype 2 | 104 | 21 | 125
  Genotype 4 | 116 | 22 | 138
  Genotype 5 | 35 | 0 | 35
  Genotype 6 | 41 | 8 | 49
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 186 | 36 | 222
    CT | 339 | 53 | 392
    TT | 94 | 26 | 120
    Missing | 5 | 1 | 6
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.3 (0.66) | 6.3 (0.58) | 6.3 (0.65)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 163 | 29 | 192
  ≥ 800,000 IU/mL | 461 | 87 | 548

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants randomized or enrolled into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | Placebo
Number analyzed (Participants) | 624 | 116
percentage of participants | 99.0 [97.9 to 99.6] | 0 [0.0 to 3.1]
Statistical Analysis 1: Comparison: SOF/VEL; Test type: Superiority or Other; p < 0.001, Binomial test — Participants in the SOF/VEL group were compared to the performance goal of 85% using a 2-sided exact 1-sample binomial test at the 0.05 significance level

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL | Placebo
Number analyzed (Participants) | 624 | 116
percentage of participants | 0.2 | 1.7

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | Placebo
Number analyzed (Participants) | 624 | 116
percentage of participants
  SVR4 | 99.2 [98.1 to 99.7] | 0 [0.0 to 3.1]
  SVR24 | 99.0 [97.9 to 99.6] | 0 [0.0 to 3.1]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Weeks 1, 2, 4, 6, 8, 10, and 12
Time Frame: Weeks 1, 2, 4, 6, 8, 10, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | Placebo
Number analyzed (Participants) | 624 | 116
percentage of participants
  Week 1 (SOF/VEL: N = 624; Placebo: N = 116) | 18.8 [15.8 to 22.0] | 0 [0.0 to 3.1]
  Week 2 (SOF/VEL: N = 624; Placebo: N = 116) | 56.9 [52.9 to 60.8] | 0 [0.0 to 3.1]
  Week 4 (SOF/VEL: N = 623; Placebo: N = 116) | 90.5 [88.0 to 92.7] | 0 [0.0 to 3.1]
  Week 6 (SOF/VEL: N = 623; Placebo: N = 115) | 98.9 [97.7 to 99.5] | 0 [0.0 to 3.2]
  Week 8 (SOF/VEL: N = 622; Placebo: N = 114) | 99.7 [98.8 to 100.0] | 0 [0.0 to 3.2]
  Week 10 (SOF/VEL: N = 622; Placebo: N = 114) | 100.0 [99.4 to 100.0] | 0 [0.0 to 3.2]
  Week 12 (SOF/VEL: N = 622; Placebo: N = 113) | 100.0 [99.4 to 100.0] | 0 [0.0 to 3.2]

5. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 1, 2, 4, 6, 8, 10, and 12
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 10, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | Placebo
Number analyzed (Participants) | 624 | 116
log10 IU/mL
  Change at Wk 1 (SOF/VEL: N= 617; Placebo: N= 114) | -4.29 (0.647) | -0.05 (0.561)
  Change at Wk 2 (SOF/VEL: N= 622; Placebo: N= 116) | -4.82 (0.685) | 0.01 (0.280)
  Change at Wk 4 (SOF/VEL: N= 617; Placebo: N= 114) | -5.08 (0.656) | -0.01 (0.297)
  Change at Wk 6 (SOF/VEL: N= 623; Placebo: N= 115) | -5.11 (0.664) | 0.07 (0.298)
  Change at Wk 8 (SOF/VEL: N= 622; Placebo: N= 113) | -5.11 (0.664) | 0.05 (0.281)
  Change at Wk 10 (SOF/VEL: N= 622; Placebo: N= 112) | -5.12 (0.662) | 0.05 (0.337)
  Change at Wk 12 (SOF/VEL: N= 622; Placebo: N= 111) | -5.12 (0.662) | -0.06 (0.580)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL | Placebo
Number analyzed (Participants) | 624 | 116
percentage of participants | 0.3 | 100

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF/VEL | Placebo
Serious Adverse Events (participants affected / at risk) | 15/624 | 0/116
Other Adverse Events (participants affected / at risk) | 393/624 | 77/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=624) | Placebo (N=116)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=624) | Placebo (N=116)
Diarrhoea (Gastrointestinal disorders) | 48 | 8
Nausea (Gastrointestinal disorders) | 75 | 13
Asthenia (General disorders) | 42 | 9
Fatigue (General disorders) | 127 | 24
Nasopharyngitis (Infections and infestations) | 80 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 6
Headache (Nervous system disorders) | 182 | 33
Insomnia (Psychiatric disorders) | 50 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years